CLINICAL TRIAL: NCT04285346
Title: A Phase 2 Open-label 12-Week Trial of Adjunctive Ganaxolone Treatment (Part A) in Tuberous Sclerosis Complex-related Epilepsy Followed by Long-term Treatment (Part B)
Brief Title: Adjunctive Ganaxolone Treatment (Part A) in TSC Followed by Long-term Treatment (Part B)
Acronym: TSC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Marinus Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1042-TSC-2001
Record Dates: First submitted 2020-02-18; First posted 2020-02-26 (Actual); Results first posted 2023-04-04 (Actual); Last update posted 2023-04-04 (Actual); Status verified 2023-03

CONDITIONS: Tuberous Sclerosis
MeSH Terms: conditions — Tuberous Sclerosis | interventions — ganaxolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Open-label (Other): ganaxolone suspension (50 mg/ml) TID for 12 weeks with 24 week extension
  Interventions: Drug: Ganaxolone

INTERVENTIONS:
Drug: Ganaxolone — titration followed by maintenance and extension period

SUMMARY:
To assess preliminary safety and efficacy of ganaxolone as adjunctive therapy for the treatment of primary seizure types in patients with genetically- or clinically-confirmed TSC-related epilepsy through the end of the 12 week treatment period.

DETAILED DESCRIPTION:
This is an OL proof of concept study of adjunctive GNX treatment in patients with a confirmed clinical diagnosis of TSC and/or a mutation in either the TSC1 or TSC2 gene. The trial consists of two parts: Part A consists of a 4-week baseline period followed by a 12-week treatment period (4-week titration and 8-week maintenance). For patients not continuing in the 24-week OLE period (Part B), a 2-week taper period followed by a 2-week safety period would follow. The main difference between Part A and Part B is the length of treatment, less frequent assessments, and the ability to alter drug doses (both GNX and other antiepileptic drug [AED] treatments which includes initiating and stopping other medications) based on investigator evaluation of the patient's clinical course during Part B. Patients with a seizure frequency reduction during the 12-week treatment period in Part A compared to baseline may continue into Part B ("OLE eligible"), to assess long-term safety, efficacy and tolerability in patients with TSC-related Epilepsy.

ELIGIBILITY:
Inclusion Criteria (Part A):

* Clinical or mutational diagnosis of TSC
* Failure to control seizures despite appropriate trial of 2 or more ASMs at therapeutic doses.
* Have at least 8 countable/witnessed primary seizures during the 4-week baseline period with at least 1 primary seizure occurring in at least 3 of the 4 weeks of baseline.

Inclusion Criteria (Part B)

• Patients have experienced ≥ 35% reduction in primary seizure frequency during the Part A treatment period compared to the 4-week Baseline Period.

Exclusion Criteria (Part A):

* Previous exposure to GNX
* Pregnant or breastfeeding
* Concurrent use of strong inducers or inhibitors of cytochrome P450 (CYP)3A4/5/7. Any strong inhibitor or inducer of CYP3A4/5/7 must be discontinued at least 28 days before Visit 2, study drug initiation. This does not include approved ASMs.
* Patients who have been taking felbamate for less than 1 year prior to screening
* Patients who test positive for tetrahydrocannabinol (THC) or non-approved cannabidiol (CBD) via plasma drug screen
* Chronic use of oral steroid medications, ketoconazole (except for topical formulations), St. John's Wort, or other IPs is not permitted
* Have an active CNS infection, demyelinating disease, degenerative neurological disease, or CNS disease deemed progressive. This includes tumor growth which in the opinion of the investigator could affect primary seizure control
* Patients with significant renal insufficiency, estimated glomerular filtration rate (eGFR) < 30 mL/min (calculated using the Cockcroft-Gault formula or Pediatric GFR calculator or Bedside Schwartz), will be excluded from study entry or will be discontinued if the criterion is met post baseline
* Have been exposed to any other investigational drug within 30 days or fewer than 5 half lives (whichever is shorter) prior to the screening visit

Ages: 2 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2020-04-08 (Actual); Primary Completion 2021-06-25 (Actual); Study Completion 2022-08-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Marinus Research Site, Los Angeles, California
  - Marinus Research Site, Palo Alto, California
  - Marinus Research Site, Boston, Massachusetts
  - Marinus Research Site, Livingston, New Jersey
  - Marinus Research Site, Durham, North Carolina
  - Marinus Research Site, Cincinnati, Ohio
  - Marinus Research Site, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was an open label proof of concept study of adjunctive Ganaxolone treatment in participants with a confirmed clinical diagnosis of Tuberous Sclerosis Complex (TSC). The trial consisted of two parts: 12-Week Treatment period and an open label extension period.
Pre-assignment Details: A total of 23 participants were enrolled in the study.
Groups:
- Treatment Period: Ganaxolone: Participants >28 kilograms (kg) were administered with Ganaxolone 1800 milligrams per day (mg/day). Following the Treatment period, participants with a seizure reduction of >=35 percent compared to the Baseline period and who did not have any other contraindications continued to be treated with Ganaxolone in the Open label period.
- Open Label: Ganaxolone: Following the Treatment period, participants with a seizure reduction of >=35 percent compared to the Baseline period and who did not have any other contraindications continued to be treated with Ganaxolone in the Open label period.
Period: Treatment Period (Up to 12 Weeks)
Arm/Group | Treatment Period: Ganaxolone | Open Label: Ganaxolone
Started | 23 | 0
Completed | 17 | 0
Not Completed | 6 | 0
Not completed — Adverse Event | 4 | 0
Not completed — Lack of Efficacy | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Period: Open Label Period (Week 12 to 38)
Arm/Group | Treatment Period: Ganaxolone | Open Label: Ganaxolone
Started | 0 | 9
Completed | 0 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety Population comprised of all participants who have received at least one dose of Ganaxolone.
Groups:
- Treatment Period: Ganaxolone: Participants >28 kg were administered with Ganaxolone 1800 milligrams per day (mg/day). Following the Treatment period, participants with a seizure reduction of >=35 percent compared to the Baseline period and who did not have any other contraindications continued to be treated with Ganaxolone in the Open label extension period.
Arm/Group | Treatment Period: Ganaxolone
Number analyzed (Participants) | 23
Age, Continuous [Mean (Standard Deviation); unit: Years] | 13.7 (8.86)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 21
  Unknown or Not Reported | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 3
  White | 17
  Declined to answer | 1
  Other-Unspecified | 2

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in 28-day Seizure Frequency Through the End of 12-Week Treatment Period
Description: Primary seizures include atonic/drop, bilateral clonic, bilateral tonic, focal motor without impairment of consciousness or awareness, focal (motor or non-motor) with impairment of consciousness or awareness, focal to bilateral tonic-clonic, generalized tonic-clonic. Baseline 28-day seizure frequency was calculated as the total number of primary seizures in the Baseline period divided by the number of days with non-missing seizure data in the Baseline period, multiplied by 28. The Baseline Visit was defined as Week 0. Percent change from Baseline in 28-day seizure frequent was calculated as the difference in post-Baseline 28-day seizure frequency and Baseline 28-day seizure frequency, divided by Baseline 28-day seizure frequency, multiplied by 100.
Time Frame: Baseline and Up to Week 12
Population: Intention to Treat (ITT) Population comprised of all participants who received at least one dose of Ganaxolone and have at least one post-Baseline efficacy assessment.
Measure: Median (95% Confidence Interval); unit: Percent change
Arm/Group | Treatment Period: Ganaxolone
Number analyzed (Participants) | 23
Percent change | -16.61 [-56.40 to 14.86]

2. Secondary Outcome: Percentage of Participants Experiencing a >=50 Percent Reduction in 28-day Primary Seizure Frequency Through the End of the 12-week Treatment Period Compared to the Baseline Period
Description: Primary seizures include atonic/drop, bilateral clonic, bilateral tonic, focal motor without impairment of consciousness or awareness, focal (motor or non-motor) with impairment of consciousness or awareness, focal to bilateral tonic-clonic, generalized tonic-clonic. Percentage of participants reporting >=50 percent reduction in seizure frequency has been presented.
Time Frame: Baseline and up to 12 Weeks
Population: ITT Population.
Measure: Number; unit: Percentage of participants
Arm/Group | Treatment Period: Ganaxolone
Number analyzed (Participants) | 23
Percentage of participants | 30.4

ADVERSE EVENTS:
Time Frame: Up to Week 12 in Treatment period and From Week 12 to Week 38 in Open label period.
Description: Safety population comprised of all participants who received at least one dose of Ganaxolone.
Groups:
- Open Label: Ganaxolone: Following the Treatment period, participants with a seizure reduction of >=35 percent compared to the Baseline period and who did not have any other contraindications continued to be treated with Ganaxolone in the Open label extension period.
Arm/Group | Treatment Period: Ganaxolone | Open Label: Ganaxolone
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/9
Serious Adverse Events (participants affected / at risk) | 3/23 | 1/9
Other Adverse Events (participants affected / at risk) | 20/23 | 3/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Period: Ganaxolone (N=23) | Open Label: Ganaxolone (N=9)
Seizure (Nervous system disorders) | 1 (1) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Angioedema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Thalamic infarction (Nervous system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Period: Ganaxolone (N=23) | Open Label: Ganaxolone (N=9)
Somnolence (Nervous system disorders) | 10 (13) | 0 (0)
Sedation (Nervous system disorders) | 3 (3) | 0 (0)
Dizziness (Nervous system disorders) | 2 (2) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 0 (0)
Ataxia (Nervous system disorders) | 1 (1) | 0 (0)
Balance disorder (Nervous system disorders) | 1 (1) | 0 (0)
Coordination abnormal (Nervous system disorders) | 1 (1) | 0 (0)
Hydrocephalus (Nervous system disorders) | 1 (1) | 0 (0)
Insomnia (Nervous system disorders) | 1 (1) | 0 (0)
Lethargy (Nervous system disorders) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 3 (3) | 0 (0)
Asthenia (General disorders) | 2 (3) | 0 (0)
Gait disturbance (General disorders) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Ear infection (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0)
Viral infection (Infections and infestations) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (1) | 0 (0)
Lip dry (Gastrointestinal disorders) | 1 (1) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Burns second degree (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Skin wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tooth fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Abnormal behaviour (Psychiatric disorders) | 1 (1) | 0 (0)
Aggression (Psychiatric disorders) | 1 (1) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Diplopia (Eye disorders) | 1 (1) | 0 (0)
Immunosuppressant drug level increased (Investigations) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-06-14): https://cdn.clinicaltrials.gov/large-docs/46/NCT04285346/Prot_000.pdf
  • Statistical Analysis Plan (2021-03-22): https://cdn.clinicaltrials.gov/large-docs/46/NCT04285346/SAP_001.pdf